CLINICAL TRIAL: NCT01905943
Title: A Multicenter, Open-Label, Single-Arm, Phase IIIb, International Study Evaluating the Safety of Obinutuzumab Alone or in Combination With Chemotherapy in Patients With Previously Untreated or Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: A Safety and Efficacy Study of Obinutuzumab Alone or in Combination With Chemotherapy in Participants With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO28543; 2013-000087-29 (EudraCT Number)
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Chlorambucil; Cyclophosphamide; fludarabine; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab (Experimental): Participants will receive obinutuzumab either alone as single agent or in combination with chemotherapy (Fludarabine/Cyclophosphamide [FC], Bendamustine or Chlorambucil) at the investigator's discretion. Each cycle is of 28-days duration.
  Interventions: Drug: Bendamustine; Drug: Chlorambucil; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine: 90 milligram per millilitre square (mg/m^2) IV over 60 minutes once daily (QD) Day 1-2 in participants previously untreated or 70 mg/m^2 I.V. over 60 minutes QD Day 1-2 in participants with relapsed/refractory disease. In non-fit participants only, investigators may opt at their own discretion to use lower initial doses of bendamustine, i.e., bendamustine 70 mg/m^2 in previously untreated participants, and bendamustine 50 mg/m^2 in relapsed/refractory subjects (over 60 minutes qd Day 1-2 for each administration).
Drug: Chlorambucil — Chlorambucil 0.5 mg/kg p.o. qd on Day 1 and Day 15 in non-fit participants only.
Drug: Cyclophosphamide — Cyclophosphamide 250 mg/m^2 I.V. over 15-30 minutes qd Day 1-3 or Cyclophosphamide 250 mg/m^2 p.o. QD Day 1-3 in fit participants only.
Drug: Fludarabine — Fludarabine 25 mg/m^2 I.V. over 30 minutes QD Day 1-3 or Fludarabine 40 mg/m^2 per os (p.o.) QD Day 1-3 in fit participants only.
Drug: Obinutuzumab — Participants will receive obinutuzumab 1000 mg IV infusion on Days 1/2 (dose split over 2 consecutive days; 100 mg on Day 1 and 900 mg on Day 2), 8 and 15 of cycle 1, and on Day 1 of Cycles 2, 3, 4, 5, and 6. Each cycle is of 28-days duration.
  Other Names: Gazyva®, RO5072759

SUMMARY:
This multicenter, open-label, single-arm study will evaluate the safety and efficacy of obinutuzumab alone or in combination with chemotherapy in participants with previously untreated or relapsed/refractory chronic lymphocytic leukemia (CLL). This is a Post-Authorization Safety Study. Participants will receive 6 cycles of single-agent obinutuzumab or obinutuzumab in combination with chemotherapy at the investigator's discretion. Each participant will be followed until 30 months after the last participant has been enrolled. Total length of the study is anticipated to be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated documented CLL according to National Cancer Institute/international workshop on CLL (NCI/iwCLL) criteria OR relapsed and/or refractory documented CLL participants requiring treatment according to NCI/iwCLL criteria; participants with up to 3 relapses are eligible
* Refractory participants if last treatment was with single-agent therapy, single-agent chemotherapy, or single-agent antibody
* Participants with 17p-deletion and/or p53 mutation may be included at the investigator's discretion
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy greater than (>) 6 months according to the investigator's opinion
* Adequate hematological function

Exclusion Criteria:

* Participants who have received more than 3 previous CLL treatment lines
* Documented transformation of CLL to aggressive lymphoma (Richter's transformation)
* Participants who are refractory to immunochemotherapy
* Participants with abnormal laboratory values
* One or more individual organ/system impairment score of 4 as assessed by the cumulative illness rating scale (CIRS) definition, excluding the eyes, ears, nose, throat and larynx organ systems
* Participants with a history of progressive multifocal leukoencephalopathy (PML)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known hypersensitivity to the study drugs
* History of prior malignancy unless the malignancy has been treated with a curative intent and in remission without treatment for greater than or equal to (>/=) 5 years prior to enrollment and with the exception of curatively-treated basal cell carcinoma, squamous cell carcinoma of the skin, low grade in situ carcinoma of the cervix, or low grade, early stage localized prostate cancer treated surgically with curative intent
* Regular treatment with corticosteroids during the 28 days prior to the start of Cycle 1, Day 1, unless administered for indications other than CLL at a dose equivalent to less than or equal to (</=) 30 milligrams per day (mg/day) prednisone
* Regular treatment with immunosuppressive medications following previous organ transplantation
* Evidence of significant, uncontrolled concomitant diseases
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of the nail beds) or a major episode of infection requiring treatment with intravenous (IV) antibiotics or hospitalization within 28 days prior to the start of Cycle 1, Day 1
* Vaccination with live vaccines within 28 days prior to start of Cycle 1, Day 1
* Major surgery (within 28 days prior to the start of Cycle 1, Day 1), other than for diagnosis
* Positive for chronic hepatitis B, hepatitis C, human T-lymphotropic virus 1 (HTLV 1) or human immunodeficiency virus (HIV) infection
* Pregnant or lactating women
* Fertile men or women of childbearing potential
* Participation in another clinical trial with drug intervention within 28 days prior to start of Cycle 1, Day 1 and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (174):
- Hospital Iturraspe, Santa Fé, Argentina
- Belgium (5):
  - Hospital Erasme; Neurologie, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - CHU Sart-Tilman, Liège
  - Sint Augustinus Wilrijk, Wilrijk
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Clinic for Internal Disease, Hematology Dept, Banja Luka
  - University Clinical Center Sarajevo, Clinic for Hematology, Sarajevo
- Brazil (8):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
  - Hospital Sirio Libanes; Centro de Oncologia, São Paulo, São Paulo
  - Hospital Estadual do Servidor Publico; Hematologia, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP; Hematologia, São Paulo, São Paulo
  - Hospital Santa Marcelina;Oncologia, São Paulo, São Paulo
- Canada (9):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Regional health authority A vitalite health network, Moncton, New Brunswick
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre; c/o Oncology Clinical Trials, Barrie, Ontario
  - Hopital Charles Lemoyne; Centre Integre de Lutte Contre Le Cancer de La Monteregie, Greenfield Park, Quebec
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - Centre de sante et de services sociaux Rimouski Neigette, Rimouski, Quebec
  - Saskatoon Cancer Centre; Uni of Saskatoon Campus, Saskatoon, Saskatchewan
  - CHU de Quebec - Hopital de l'Enfant-Jesus; Unite de Recherche en Hematologie et Oncologie, Québec
- Egypt (2):
  - Cairo University Hospital Al Kasr El Ainy, Cairo
  - National Cancer Institute, Cairo
- Estonia (2):
  - North Estonia Regional Hospital; Hematology, Tallinn
  - Tartu Uni Hospital; Hematology - Oncology Clinic, Tartu
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital; Hematology, Tampere
  - Turku Uni Central Hospital; Dept of Internal Medicine, Turku
- France (25):
  - Hotel Dieu; Medecine D, Angers
  - Ch Victor Dupouy; Hematologie, Argenteuil
  - Hopital Augustin Morvan; Hematologie, Brest
  - Hopital Cote De Nacre; Hematologie Biologique, Caen
  - Chu Estaing; Hematologie Clinique Adultes, Clermont-Ferrand
  - Hopital Henri Mondor; Hematologie Clinique, Créteil
  - Chu Site Du Bocage;Hematologie Clinique, Dijon
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Ch Du Mans; Medecine Hematologie Oncologie, Le Mans
  - Hopital Claude Huriez; Hematologie, Lille
  - Hopital Uni Ire Dupuytren; Hematologie, Limoges
  - Hopital Saint Eloi; Hematologie Oncologie Medicale, Montpellier
  - Hopital Emile Muller; Hematologie, Mulhouse
  - Hopital Hotel Dieu Et Hme;Hopital De Jour, Nantes
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - Hopital Saint Antoine; Hematologie Clinique, Paris
  - Hopital Pitie Salpetriere; Hematologie Clinique, Paris
  - Hopital Saint Jean; Hematologie, Perpignan
  - Hopital De Haut Leveque; Hematologie Clinique, Pessac
  - Ch Lyon Sud; Hemato Secteur Jules Courmont, Pierre-Bénite
  - Centre Hospitalier René Dubos; Hematologie, Pontoise
  - Hopital Robert Debre; Hematologie Clinique, Reims
  - Centre Henri Becquerel; Hematologie, Rouen
  - Centre Hospitalier de Saint Brieuc - Hôpital Yves Le Foll, Saint-Brieuc
  - Hopital Bretonneau; Hematologie Therapie Cellulaire, Tours
- Germany (16):
  - Hämatologisch-onkologische Praxis Dr. med. - Heinrich, - Bangerter, Augsburg
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Onkologisches Zentrum am Bethanien-Kankenhaus, Frankfurt
  - Gemeinschaftspraxis; Prof. Dr. Michael Kiehl und Dr.med. Wolfgang Stein, Frankfurt (Oder)
  - Dres.Andreas Ammon und Dirk Meyer, Göttingen
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
  - Onkologische Gemeinschaftspraxis, Magdeburg
  - Kliniken Ostalb, Stauferklinikum Schwäbisch-Gmünd; Zentrum für Innere Medizin, Mutlangen
  - Dres. Hans-Dieter Schick Dorothea Schick Burkhard Schmidt u.w., München
  - Gemeinschaftspraxis Dr. med. Holger Klaproth / Dr. med. Anca Astrid Cura, Neunkirchen/Saar
  - eps - early phase GmbH, Pößneck
  - Oncologianova GmbH - Gesellschaft für Innovationen in der Onkologie, Recklinghausen
  - Schwerpunktpraxis & Tagesklinik f. Hämatologie & Onkologie Regensdorf / Schwandorf / Wörth, Regensburg
  - Universitätsklinikum Ulm; Medizinische Uni-Klinik III Abt. Innere Medizin III Hämatologie u. Onkolo., Ulm
  - Onkologische Schwerpunktpraxis Dres. Rudolf Schlag und Björn Schöttker, Würzburg
- Greece (5):
  - General Hospital of Athens Evangelismos; Hematology, Athens
  - Laiko General Hospital of Athens; A Propedeutical Clinic of Internal Medicine, Athens
  - Laiko General Hospital; Hematology Clinic, Athens
  - University Hospital of Ioannina; Hematology, Ioannina
  - Georgios Papanikolaou Hospital; Hematology Department, Thessaloniki
- Ireland (3):
  - Mater Misericordiae Uni Hospital; Oncology, Dublin
  - University Hospital Limerick - Oncology, Limerick
  - Waterford Regional Hospital; Department Of Medical Oncology, Waterford
- Israel (5):
  - Soroka Medical Center; Hematology Deptartment, Beersheba
  - Bnei-Zion Medical Center; Hematology Dept, Haifa
  - Hadassah Ein Karem Hospital; Haematology, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Ichilov Sourasky Medical Center; Heamatology, Tel Aviv
- Italy (18):
  - Azienda ospedaliera oo rr di foggi; Hematology, Foggia, Apulia
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - Az. Osp. Pugliese; Divisione de Ematologia, Catanzaro, Calabria
  - Ospedale Cardarelli; Divisione Di Ematologia, Napoli, Campania
  - Arcispedale S. Anna; Sezione Di Ematologia, Ferrara, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - AUSL di Piacenza - Ospedale "Guglielmo da Saliceto";U.O. Ematologia, Piacenza, Emilia-Romagna
  - Az. Osp. S. Maria Delle Croci; U.O. Di Ematologia, Ravenna, Emilia-Romagna
  - Ospedale Infermi Di Rimini; Unità Operativa di Oncologia e Oncoematologia, Rimini, Emilia-Romagna
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia; Dip Biot Cel e Ematol, Rome, Lazio
  - Uni Degli Studi Di Genova; 1A Divisione Di Ematologia, Genoa, Liguria
  - Ospedale Maggiore Di Milano; U.O. Ematologia I - Padiglione Marcora, Milan, Lombardy
  - ASST GRANDE OSPEDALE METROPOLITANO NIGUARDA; Struttura Complessa di Ematologia, Milan, Lombardy
  - Univ. Piemonte Est Amedeo Avogadro; Div.Ematologia- Dip.Clinica Med.Sperim.& Ircad, Novara, Piedmont
  - Ospedale Molinette - Universita' Di Torino; Cliniche Universitarie Ematologia I, Turin, Piedmont
  - Ospedale Oncologico A Businco-Cagliari; Ematologia Sez., Cagliari, Sardinia
  - Azienda USL 6 Livorno - P.O. Livorno; U.O. Ematologia Clinica, Livorno, Tuscany
- RECUH, Oncology Centre of Latvia; Clinic of Chemotherapy and Heamatology, Riga, Latvia
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Clinic, Hematology, Oncology and Tranfusion Medicine Center, Vilnius
- Mexico (5):
  - Hospital General De Culiacan; Servicio De Hematologia, Culiacán
  - Hospital General de México; Haematology, Mexico City
  - Centro Medico Nacional Sxxi - Imss; Haematology, Mexico City
  - Hospital Universitario Dr. Jose E. Gonzalez; Haematology, Monterrey
  - Centro de Estudios Clinicos de Queretaro (CECLIQ), Querétaro
- University Clinic of Hematology Skopje, Hospital Care Department, Skopje, North Macedonia
- Poland (4):
  - Katedra i Klinika Hematoonkologii i Transplantacji Szpiku; Uniwersytetu Medycznego w Lublinie, Lublin
  - Oddzial Kliniczny Hematologii SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Szpital Wojewodzki w Opolu, Oddzial Hematologii i Onkologii Hematologicznej, Opole
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka; Oddział Chorób Wewnetrznych/Hematologiczny, Słupsk
- Portugal (2):
  - Hospital de Santa Maria; Servico de Hematologia e Transplantacao de Medula, Lisbon
  - IPO do Porto; Servico de Onco-Hematologia, Porto
- Romania (4):
  - Policlinica de Diagnostic Rapid, Brasov
  - Spitalul Clinic Judetean de Urgenta Brasov; Clinica de Hematologie, Brasov
  - Spitalul Clinic Coltea; Clinica de Hematologie, Bucharest
  - Spitalul Clinic municipal de Urgenta Timisoara; Clinica de Hematologie, Timișoara
- Russia (4):
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow
  - Vladimirskiy Regional Scientific Research Inst. ; Hematology, Moscow
  - Almazov Federal Heart, Blood and Endocrinilogy Centre; Hematology department, Saint Petersburg
  - Regional Oncology Center, Volgograd
- Institute of Hematology, Belgrade, Serbia
- Slovakia (2):
  - Fakultna Nemocnica Roosevelta; Dept. of Haematology, Banská Bystrica
  - National Oncology Inst. ; Dept. of Haematology, Bratislava
- Slovenia (3):
  - Hospital Celje; Haematology Dept, Celje
  - Clinical Center Ljubljana; Haematology Dept, Ljubljana
  - Hospital Maribor; Haematology Dept, Maribor
- South Korea (3):
  - Pusan University Hospital, Busan
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
- Spain (12):
  - Hospital De Txagorritxu; Servicio de Hematologia, Vitoria-Gasteiz, Alava
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Hematologia, Badalona, Barcelona
  - Complejo Hospitalario San Millan - San Pedro; Servicio Hematologia, Logroño, La Rioja
  - Hospital Quiron de Madrid; Servicio de Hematologia, Pozuelo de Alarcón, Madrid
  - Hospital San Pedro De Alcantara; Servicio de Hematologia, Cáceres
  - Hospital Universitario Reina Sofia; Servicio de Hematologia, Córdoba
  - Hospital Infanta Leonor; Servicio de Hematologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Hematología, Madrid
  - Complejo Hospitalario Universitario de Ourense, Servicio de Hematologia, Ourense
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- Sweden (4):
  - Universitetssjukhuset i Linköping, Hematologkliniken, Linköping
  - Skane University Hospital Malmo/Lund, Dept.of Hematology and Coagulation Disorders, Malmo
  - Uddevalla Sjukhus; Medicinkliniken, Uddevalla
  - Akademiska Sjukhuset, Uppsala
- Switzerland (7):
  - Kantonsspital Aarau; Zentrum Für Onkologie, Hämatologie & Transfusionsmedizin, Aarau
  - Universitätsspital Basel; Hämatologie, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
  - HUG; Hématologie, Geneva
  - Luzerner Kantonsspital, Hämatologie, Lucerne
  - OnkoZentrum Zuerich, Zurich
- Thailand (5):
  - King Chulalongkorn Memorial Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Ramathibodi Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Siriraj Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Chiang Mai Uni Hospital; Division of Hematology,Dept of Medicine,Faculty of Medicine, Chiang Mai
  - Srinagarind Hospital, Khon Kaen Uni ; Dept of Medicine, Khon Kaen
- Turkey (Türkiye) (10):
  - Cukurova Uni ; Hematology, Adana
  - Ankara Numune Egitim Ve Arastirma Hastanesi; Hematoloji Klinigi, Ankara
  - Ankara University; Hematology, Ankara
  - Pamukkale Uni. Med. Fac., Denizli
  - Gaziantep University Medical School; Hematology, Gaziantep
  - Istanbul Uni Capa Hospital; Hematology, Istanbul
  - Dokuz Eylul Uni ; Hematology, Izmir
  - Erciyes Uni ; Hematology, Kayseri
  - Ondokuzmayis University Medical Faculty Heamatology Department, Samsun
  - Karadeniz Technical Uni School of Medicine; Hematology, Trabzon

REFERENCES:
- [Derived] Stilgenbauer S, Bosch F, Ilhan O, Kisro J, Mahe B, Mikuskova E, Osmanov D, Reda G, Robinson S, Tausch E, Turgut M, Wojtowicz M, Bottcher S, Perretti T, Trask P, Van Hoef M, Leblond V, Foa R. Safety and efficacy of obinutuzumab alone or with chemotherapy in previously untreated or relapsed/refractory chronic lymphocytic leukaemia patients: Final analysis of the Phase IIIb GREEN study. Br J Haematol. 2021 Apr;193(2):325-338. doi: 10.1111/bjh.17326. Epub 2021 Feb 19. PMID 33605445
- [Derived] Bosch F, Cantin G, Cortelezzi A, Knauf W, Tiab M, Turgut M, Zaritskey A, Merot JL, Tausch E, Trunzer K, Robson S, Gresko E, Bottcher S, Foa R, Stilgenbauer S, Leblond V. Obinutuzumab plus fludarabine and cyclophosphamide in previously untreated, fit patients with chronic lymphocytic leukemia: a subgroup analysis of the GREEN study. Leukemia. 2020 Feb;34(2):441-450. doi: 10.1038/s41375-019-0554-1. Epub 2019 Aug 27. PMID 31455851
- [Derived] Stilgenbauer S, Leblond V, Foa R, Bottcher S, Ilhan O, Knauf W, Mikuskova E, Renner C, Tausch E, Woszczyk D, Gresko E, Lundberg L, Moore T, Morris T, Robson S, Bosch F. Obinutuzumab plus bendamustine in previously untreated patients with CLL: a subgroup analysis of the GREEN study. Leukemia. 2018 Aug;32(8):1778-1786. doi: 10.1038/s41375-018-0146-5. Epub 2018 Apr 27. PMID 29749403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 195 centers in 31 countries
Pre-assignment Details: A total of 1131 subjects were screened and 979 subjects were enrolled. Due to compliance issues a site in Romania was closed. Seven subjects were excluded from the analysis, because data integrity was impacted by the site's non-compliance. Hence, data analysis is reported for 972 enrolled subjects.
Groups:
- Obinutuzumab: Participants received obinutuzumab either alone as single agent, or in combination with chemotherapy (Fludarabine/Cyclophosphamide [FC], Bendamustine or Chlorambucil).
Period: Overall Study
Arm/Group | Obinutuzumab
Started | 972
Completed | 658 (All patients provide reason at final analysis)
Not Completed | 314
Not completed — Withdrawal of consent | 90
Not completed — Lost to Follow-up | 16
Not completed — Investigator discretion | 7
Not completed — Death | 186
Not completed — Adverse Event | 3
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all participants enrolled in the study regardless of whether or not they received any study drug.
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 972
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 355
  Male | 617

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs, including AEs of Special Interest and AEs of Particular Interest, were reported based on the national cancer institute common terminology criteria for AEs, Version 4.0 (NCI-CTCAE, v4.0). Reported are the number of subjects with AEs, Grade 3-5 AEs, and Serious Adverse Events (SAEs).
Time Frame: Baseline up to time of primary completion (3 years)
Population: The safety population was defined as all participants who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 971
Participants
  AEs | 950
  Grade 3-5 AEs | 780
  SAEs | 516

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: The following AEs were defined as AESIs: AEs with the preferred term Tumour Lysis Syndrome (TLS), Infusion-Related Reactions (IRRs) defined as AEs that occurred during or within 24 hours of the completion of obinutuzumab infusion and were assessed as related to obinutuzumab by the Investigator, Infections defined as AEs from System Organ Class (SOC) "Infections and infestations" and AEs with the preferred term Neutropenia. Reported are number of participants with total AESIs, IRRs, Infections, Neutropenia and TLS.
Time Frame: Baseline up to time of primary completion (3 years)
Population: The safety population was defined as all participants who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 971
Participants
  Total AESIs | 905
  IRRs | 635
  Neutropenia | 599
  Infections | 521
  TLS | 62

3. Primary Outcome: Number of Participants With Adverse Events of Particular Interest (AEPIs)
Description: The following AEs were defined as AEPIs: AEs with the preferred term Progressive multifocal leukoencephalopathy (PML), hepatitis B reactivation defined as AEs with preferred term containing "Hepatitis B" or "hepatitis acute", thrombocytopenia defined via Roche MedDRA basket subgroup "haematopoietic thrombocytopenia", second malignancies defined as AEs from the SOC "Neoplasms benign, malignant and unspecified" starting 6 months after the first study drug intake, second malignancies based on standardised MedDRA queries (SMQ) starting 6 months after the first study drug intake based on the MedDRA SMQ "Malignant or unspecified tumours", in which benign neoplasms are not included, Cardiac events including AEs from the SOC "Cardiac disorders", and hemorrhagic events defined via Roche MedDRA basket subgroup "Haemorrhagic events". Reported are number of participants with total AEPIs and each of the AEPI categories.
Time Frame: Baseline up to time of primary completion (3 years)
Population: The safety population was defined as all participants who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 971
Participants
  Total AEPIs | 467
  Thrombocytopenia | 314
  Cardiac events | 109
  Second malignancies | 82
  Second malignancies (SMQ) | 75
  Hemorrhagic events | 69
  Hepatitis B reactivation | 3
  PML | 1

4. Secondary Outcome: Percentage of Participants With Overall Response (OR) at Final Response Assessment (FRA)
Description: OR: percentage of participants with complete response (CR) or CR with incomplete marrow recovery (CRi), or partial response (PR), as determined by the investigator based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) tumor response criteria. CR: Peripheral blood lymphocytes 4,000/mcL, no significant lymphadenopathy, no hepatomegaly and splenomegaly, no disease symptoms, blood counts: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L and bone marrow normocellular for age. Cri: CR with persistent cytopenia. PR: >/= 50% decrease in peripheral blood lymphocyte count AND >/= 50% reduction in lymphadenopathy OR >/= 50% reduction of liver enlargement OR >/= 50% reduction of spleen PLUS one of the following: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L OR >/= 50% increase in neutrophils, platelets or hemoglobin.
Time Frame: 3 months after the last dose of study treatment (up to approximately 5 years)
Population: The ITT population was defined as all participants enrolled in the study regardless of whether or not they received any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- G Mono: Previously Untreated Fit: Participants with obinutuzumab monotherapy who were previously untreated fit. Fit participants were defined as having a total Cumulative Illness Rating Scale (CIRS) score ≤6 and creatinine clearance (CrCl) ≥70 mL/min.
- G Mono: Previously Untreated Unfit: Participants with obinutuzumab monotherapy who were previously untreated unfit. Non fit participants were defined as having a CIRS score >6 and/or CrCl <70 mL/min.
- G Mono: Relapsed/Refractory: Participants with obinutuzumab monotherapy who had documented relapsed/refractory chronic lymphocytic leukemia (CLL).
- G-Benda: Previously Untreated Fit: Participants with obinutuzumab in combination with bendamustine who were previously untreated fit. Fit participants were defined as having a total CIRS score <=6 and CrCl >=70 mL/min.
- G-Benda: Previously Untreated Unfit: Participants with obinutuzumab in combination with bendamustine who were previously untreated unfit. Non fit Participants were defined as having a CIRS score >6 and/or CrCl <70 mL/min.
- G-Benda: Relapsed/Refractory: Participants with obinutuzumab in combination with bendamustine who had documented relapsed/refractory chronic lymphocytic leukemia (CLL).
- G-FC: Previously Untreated Fit: Participants with obinutuzumab in combination with fludarabine and cyclophosphamide who were previously untreated fit. Fit subjects were defined as having a total CIRS score <=6 and CrCl >=70 mL/min.
- G-FC: Previously Untreated Unfit: Participants with obinutuzumab in combination with fludarabine and cyclophosphamide who were previously untreated unfit. Non fit participants were defined as having a CIRS score >6 and/or CrCl <70 mL/min. This is a Protocol deviation: unfit subjects were incorrectly assigned to the G-FC treatment regimen.
- G-FC: Relapsed/Refractory: Participants with obinutuzumab in combination with fludarabine and cyclophosphamide who had documented relapsed/refractory chronic lymphocytic leukemia (CLL). This is a Protocol deviation: 5 unfit subjects were incorrectly assigned to this relapsed/refractory G-FC treatment regimen.
- G-Clb: Previously Untreated Fit: Participants with obinutuzumab in combination with chlorambucil who were previously untreated fit. Fit participants were defined as having a total CIRS score <=6 and CrCl >=70 mL/min.
- G-Clb: Previously Untreated Unfit: Participants with obinutuzumab in combination with chlorambucil who were previously untreated unfit. Non fit participants were defined as having a CIRS score >6 and/or CrCl <70 mL/min.
- G-Clb: Relapsed/Refractory: Participants with obinutuzumab in combination with chlorambucil who had documented relapsed/refractory chronic lymphocytic leukemia (CLL).
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
percentage of participants | 71.0 [52.0 to 85.8] | 59.4 [40.6 to 76.3] | 41.5 [29.4 to 54.4] | 83.9 [77.5 to 89.1] | 81.6 [75.1 to 87.0] | 73.2 [66.3 to 79.3] | 90.0 [83.8 to 94.4] | 84.6 [54.6 to 98.1] | 85.0 [70.2 to 94.3] | 100 [2.5 to 100.0] | 82.1 [70.8 to 90.4] | 56.5 [41.1 to 71.1]

5. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD)-Negativity as Assessed by Flow Cytometry
Description: MRD-negativity was defined as the presence of less than 1 chronic lymphocytic leukemia (CLL) cell per 10,000 leukocytes in blood and bone marrow as assessed by flow cytometry 3 months after last dose of study treatment (i.e. at final response assessment [FRA] visit).
Time Frame: 3 months after the last dose of study treatment (up to approximately 5 years)
Population: The intent-to-ship (ITS) population included all participants from the ITT population whose MRD samples at the FRA could be shipped to the central laboratory within 48 hours.
Measure: Number; unit: percentage of participants
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
percentage of participants
  Blood: number analyzed (Participants) | 24 | 26 | 49 | 149 | 147 | 161 | 125 | 12 | 33 | 0 | 53 | 32
  Blood | 8.3 | 23.1 | 4.1 | 63.1 | 65.3 | 39.8 | 72.0 | 58.3 | 51.5 |  | 9.4 | 6.3
  Bone Marrow: number analyzed (Participants) | 24 | 26 | 49 | 149 | 147 | 161 | 125 | 12 | 33 | 0 | 53 | 32
  Bone Marrow | 4.2 | 3.8 | 2.0 | 31.5 | 27.2 | 14.9 | 40.0 | 41.7 | 24.2 |  | 5.7 | 3.1

6. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR)
Description: BOR was defined as the percentage of participants with the best response obtained throughout the trial with CR, CRi, or PR, as determined by the investigator based on IWCLL tumor response criteria. CR: Peripheral blood lymphocytes 4,000/mcL, no significant lymphadenopathy, no hepatomegaly and splenomegaly, no disease symptoms, blood counts: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L and bone marrow normocellular for age. Cri: CR with persistent cytopenia. PR: >/= 50% decrease in peripheral blood lymphocyte count AND >/= 50% reduction in lymphadenopathy OR >/= 50% reduction of liver enlargement OR >/= 50% reduction of spleen PLUS one of the following: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L OR >/= 50% increase in neutrophils, platelets or hemoglobin.
Time Frame: Baseline, Day 85, end of treatment or early termination, and follow-up, assessed up to disease progression or death, whichever occurs first (up to approximately 5 years)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
percentage of participants | 83.9 [66.3 to 94.5] | 71.9 [53.3 to 86.3] | 60.0 [47.1 to 72.0] | 91.7 [86.4 to 95.4] | 93.9 [89.3 to 96.9] | 86.8 [81.2 to 91.3] | 97.1 [92.8 to 99.2] | 84.6 [54.6 to 98.1] | 97.5 [86.8 to 99.9] | 100 [2.5 to 100.0] | 94.0 [85.4 to 98.3] | 84.8 [71.1 to 93.7]

7. Secondary Outcome: Median Time to Progression-Free Survival (PFS)
Description: Kaplan Meier estimate of the median PFS was defined as the time at which half of the participants have progressed (progressive disease [PD]) based on IWCLL tumor response criteria or died from any cause, whichever occurred first. PD: at least one of the following: >/= 50% increase in the absolute number of circulating lymphocytes to at least 5,000/mcL, appearance of new palpable lymph nodes, >/= 50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, >/= 50% increase in the enlargement of the liver and/or spleen, transformation to more aggressive histology, progression of any cytopenia, decrease of hemoglobin levels by more than 20 g/L or to less than 100 g/L, decrease of platelet counts by more than 50% or to less than 100,000 /mcL, decrease of neutrophil counts by more than 50% or to less than 1,000/mcL.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
months | 43.0 [17.0 to NA] — Upper limit of 95% CI could not be estimated as too few patients had an event. | 21.2 [14.9 to NA] — Upper limit of 95% CI could not be estimated as too few patients had an event. | 17.6 [12.5 to 20.0] | 58.0 [44.5 to 58.0] | NA [45.4 to NA] — Median and Upper Limit 95% CI could not be estimated as too few patients had an event. | 28.6 [24.2 to 31.1] | NA [53.7 to NA] — Median and Upper Limit 95% CI could not be estimated as too few patients had an event. | NA [19.0 to NA] — Median and Upper Limit 95% CI could not be estimated as too few patients had an event. | 24.8 [19.3 to 35.0] | 31.3 [NA to NA] — 95% CI could not be estimated as too few patients had an event. | 31.8 [27.7 to 36.4] | 14.1 [10.8 to 22.1]

8. Secondary Outcome: Median Time to Response (TTR)
Description: Kaplan Meier estimate of median TTR was defined as the time at which half of the participants reached CR or PR based on IWCLL tumor response criteria. CR: Peripheral blood lymphocytes 4,000/mcL, no significant lymphadenopathy, no hepatomegaly and splenomegaly, no disease symptoms, blood counts: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L and bone marrow normocellular for age. PR: >/= 50% decrease in peripheral blood lymphocyte count AND >/= 50% reduction in lymphadenopathy OR >/= 50% reduction of liver enlargement OR >/= 50% reduction of spleen PLUS one of the following: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L OR >/= 50% increase in neutrophils, platelets or hemoglobin.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
months | 3.6 [3.2 to 3.8] | 3.6 [3.3 to 3.9] | 3.9 [3.7 to 4.4] | 3.5 [3.4 to 3.6] | 3.5 [3.5 to 3.7] | 3.7 [3.5 to 3.7] | 3.6 [3.5 to 3.7] | 4.1 [3.3 to 7.9] | 3.6 [3.4 to 3.7] | 3.3 [NA to NA] — Lower Limit and Upper limit of 95% CI could not be estimated as too few patients had an event. | 3.6 [3.4 to 3.7] | 3.7 [3.5 to 3.8]

9. Secondary Outcome: Median Time to Event-Free Survival (EFS)
Description: Kaplan Meier estimate of median EFS is the time at which half of the participants have progressed as assessed by investigator based on IWCLL tumor response criteria, or have initiated a non-protocol-specified anti-leukemia therapy or died, whichever occurs first. PD: at least 1 of the following: >/= 50% increase in absolute number of circulating lymphocytes to at least 5,000/mcL, appearance of new palpable lymph nodes, >/= 50% increase in longest diameter of any previous site of clinically significant lymphadenopathy, >/= 50% increase in enlargement of liver and/or spleen, transformation to more aggressive histology, progression of any cytopenia, decrease of hemoglobin levels by more than 20 g/L or to less than 100 g/L, decrease of platelet counts by more than 50% or to less than 100,000 /mcL, decrease of neutrophil counts by more than 50% or to less than 1,000/mcL.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
months | 35.2 [15.6 to NA] — Upper limit of 95% CI could not be estimated as too few patients had an event. | 17.9 [14.5 to NA] — Upper limit of 95% CI could not be estimated as too few patients had an event. | 14.0 [9.1 to 17.9] | 58.0 [44.5 to 58.0] | 52.9 [44.7 to NA] — Upper limit of 95% CI could not be estimated as too few patients had an event. | 25.1 [21.0 to 30.4] | NA [53.7 to NA] — Median and Upper limit of 95% CI could not be estimated as too few patients had an event. | NA [17.8 to NA] — Median and Upper limit of 95% CI could not be estimated as too few patients had an event. | 24.2 [18.7 to 33.8] | 31.3 [NA to NA] — Lower limit and Upper limit of 95% CI could not be estimated as too few patients had an event. | 31.8 [27.7 to 36.4] | 13.7 [10.5 to 18.0]

10. Secondary Outcome: Median Time to Overall Survival (OS)
Description: Kaplan Meier estimate of median OS was defined as the time at which half of the participants had died, regardless of the cause of death.
Time Frame: Baseline until death (Approximately up to 5 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [40.7 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [42.1 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [55.3 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [35.2 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event.

11. Secondary Outcome: Median Time to New Anti-Leukemia Therapy (TTNT)
Description: Kaplan Meier estimate of median TTNT was defined as the time at which half of the participants have initiated a new anti-leukemic therapy.
Time Frame: Baseline until end of study (up to approximately 5 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
months | NA [25.0 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [27.5 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | 22.5 [14.8 to 27.0] | NA [53.5 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI Lower Limit and Upper Limit could not be estimated as too few patients had an event. | 38.3 [31.5 to 42.0] | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [35.0 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | 32.6 [28.2 to NA] — 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI Lower Limit and Upper Limit could not be estimated as too few patients had an event. | 53.7 [37.1 to NA] — 95% CI Upper Limit could not be estimated as too few patients had an event. | 20.4 [13.7 to 43.3]

12. Secondary Outcome: Median Time to Duration of Response (DoR)
Description: Kaplan Meier estimate of median DoR was defined as the time at which half of the responding (PR or CR) participants had progressed (PD) or died from any cause, whichever occurred first. PR: >/= 50% decrease in peripheral blood lymphocyte count AND >/= 50% reduction in lymphadenopathy OR >/= 50% reduction of liver enlargement OR >/= 50% reduction of spleen PLUS one of the following: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L OR >/= 50% increase in neutrophils, platelets or hemoglobin. CR: Peripheral blood lymphocytes 4,000/mcL, no significant lymphadenopathy, no hepatomegaly and splenomegaly, no disease symptoms, blood counts: neutrophils >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 110 g/L and bone marrow normocellular for age. PD: as defined in the description for Event-Free Survival outcome measure.
Time Frame: as for outcome 6
Population: The ITT population was defined as all participants enrolled in the study regardless of whether or not they received any study drug. Number of participants analyzed indicates participants who took part in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G Mono: Previously Untreated Fit | G Mono: Previously Untreated Unfit | G Mono: Relapsed/Refractory | G-Benda: Previously Untreated Fit | G-Benda: Previously Untreated Unfit | G-Benda: Relapsed/Refractory | G-FC: Previously Untreated Fit | G-FC: Previously Untreated Unfit | G-FC: Relapsed/Refractory | G-Clb: Previously Untreated Fit | G-Clb: Previously Untreated Unfit | G-Clb: Relapsed/Refractory
Number analyzed (Participants) | 31 | 32 | 65 | 168 | 179 | 190 | 140 | 13 | 40 | 1 | 67 | 46
months | 40.1 [26.3 to NA] — 95% CI Upper Limit could not be estimated as too few patients had an event. | 20.1 [12.1 to NA] — 95% CI Upper Limit could not be estimated as too few patients had an event. | 15.0 [12.1 to 19.9] | 55.0 [44.2 to 55.0] | 49.3 [44.2 to NA] — 95% CI Upper Limit could not be estimated as too few patients had an event. | 25.5 [21.2 to 29.7] | NA [50.1 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | NA [48.3 to NA] — Median and corresponding 95% CI Upper Limit could not be estimated as too few patients had an event. | 21.2 [15.1 to 32.1] | 28.1 [NA to NA] — 95% CI Lower Limit and Upper Limit could not be estimated as too few patients had an event. | 28.1 [24.3 to 34.8] | 12.3 [7.3 to 20.6]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: The safety population was defined as all participants who received at least one dose of study medication. AEs that were entered into the data base at the time of the data base lock were included in the AE analysis.
Groups:
- G-Mono: Participants received obinutuzumab alone as single agent.
- G-Benda: Participants received obinutuzumab in combination with bendamustine.
- G-FC: Participants received obinutuzumab in combination with fludarabine/cyclophosphamide (FC).
- G-Clb: Participants received obinutuzumab in combination with chlorambucil.
Arm/Group | G-Mono | G-Benda | G-FC | G-Clb
Serious Adverse Events (participants affected / at risk) | 71/127 | 335/537 | 107/193 | 66/114
Other Adverse Events (participants affected / at risk) | 108/127 | 503/537 | 184/193 | 107/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Mono (N=127) | G-Benda (N=537) | G-FC (N=193) | G-Clb (N=114)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 3 (3) | 1 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 43 (49) | 20 (25) | 3 (3)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (10) | 62 (100) | 28 (50) | 6 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 17 (17) | 6 (6) | 5 (5)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (9) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 3 (3) | 5 (5) | 0 (0) | 1 (5)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 7 (7) | 1 (1) | 4 (4)
General physical health deterioration (General disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (7) | 23 (27) | 11 (11) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Allergy to immunoglobulin therapy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (5) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (5) | 0 (0) | 2 (3)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 12 (13) | 65 (90) | 15 (16) | 17 (18)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 10 (10) | 5 (5) | 3 (4)
Septic shock (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 7 (8) | 1 (1) | 2 (3)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 4 (5) | 1 (1) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cryptosporidiosis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B Reactivation (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Infective exacerbation chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 5 (5) | 7 (7) | 2 (2)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visceral leishmaniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
West nile viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Listeriosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Retinitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation mucositis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 30 (30) | 3 (3) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fistula inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6) | 1 (1) | 2 (2)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (10) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6) | 0 (0) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 8 (10) | 1 (1) | 2 (2)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5) | 1 (1) | 1 (1)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 6 (7) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coombs Negative Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal Degeneration (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemophagocytic (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Legionella Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Respiratory (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tick-Borne Viral Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular Device Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dislocation of Vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fractured Ischium (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Steroid Diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Basosquamous Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraductal Papillary Mucinous Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral T-Cell Lymphoma Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial Rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Mono (N=127) | G-Benda (N=537) | G-FC (N=193) | G-Clb (N=114)
Anaemia (Blood and lymphatic system disorders) | 19 (28) | 134 (174) | 50 (76) | 27 (35)
Leukopenia (Blood and lymphatic system disorders) | 7 (10) | 70 (119) | 27 (45) | 8 (12)
Neutropenia (Blood and lymphatic system disorders) | 45 (130) | 288 (645) | 138 (416) | 58 (127)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (34) | 162 (253) | 67 (116) | 34 (54)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 53 (88) | 11 (19) | 2 (3)
Constipation (Gastrointestinal disorders) | 8 (10) | 72 (84) | 24 (30) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 83 (114) | 38 (44) | 11 (12)
Nausea (Gastrointestinal disorders) | 23 (27) | 144 (206) | 75 (147) | 26 (33)
Vomiting (Gastrointestinal disorders) | 9 (9) | 68 (87) | 44 (67) | 15 (16)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 24 (30) | 10 (10) | 4 (5)
Asthenia (General disorders) | 8 (9) | 48 (61) | 30 (42) | 14 (17)
Chest discomfort (General disorders) | 7 (7) | 15 (15) | 7 (7) | 3 (3)
Chills (General disorders) | 18 (19) | 92 (110) | 30 (32) | 19 (22)
Fatigue (General disorders) | 7 (7) | 71 (85) | 19 (25) | 23 (27)
Pyrexia (General disorders) | 28 (33) | 173 (247) | 61 (93) | 28 (39)
Oedema peripheral (General disorders) | 4 (5) | 31 (37) | 3 (4) | 9 (15)
Bronchitis (Infections and infestations) | 11 (12) | 39 (43) | 18 (23) | 6 (8)
Influenza (Infections and infestations) | 5 (5) | 13 (16) | 12 (12) | 5 (5)
Nasopharyngitis (Infections and infestations) | 9 (11) | 25 (28) | 19 (24) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 48 (62) | 14 (17) | 5 (7)
Urinary tract infection (Infections and infestations) | 6 (9) | 29 (35) | 7 (9) | 11 (16)
Sinusitis (Infections and infestations) | 4 (4) | 16 (18) | 14 (19) | 5 (8)
Respiratory tract infection (Infections and infestations) | 5 (6) | 12 (19) | 6 (7) | 7 (8)
Alanine aminotransferase increased (Investigations) | 4 (4) | 13 (14) | 11 (12) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 15 (15) | 10 (10) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 19 (21) | 7 (9) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 35 (37) | 13 (15) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 44 (45) | 11 (15) | 11 (12)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 33 (36) | 7 (8) | 10 (11)
Headache (Nervous system disorders) | 10 (18) | 46 (57) | 23 (25) | 10 (10)
Tremor (Nervous system disorders) | 6 (6) | 11 (11) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 3 (5) | 22 (23) | 4 (4) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 57 (70) | 28 (33) | 17 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 53 (66) | 24 (24) | 11 (13)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 21 (22) | 8 (8) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 25 (30) | 11 (11) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 46 (63) | 24 (31) | 11 (15)
Hypertension (Vascular disorders) | 7 (7) | 44 (51) | 16 (17) | 5 (5)
Hypotension (Vascular disorders) | 10 (12) | 53 (61) | 17 (20) | 16 (18)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 24 (26) | 5 (5) | 6 (6)
Pneumonia (Infections and infestations) | 4 (6) | 28 (33) | 9 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.